CLINICAL TRIAL: NCT02977208
Title: Impact of Genetic Polymorphisms of OCT2 and OCTN1 on the Kinetic Disposition of Gabapentin in Patients Undergoing Chronic Use of the Drug
Brief Title: Impact of Polymorphisms of OCT2 and OCTN1 on the Kinetic Disposition of Gabapentin in Patients Undergoing Chronic Use
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: São Paulo State University (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Priscila Akemi Yamamoto, Principal investigator, São Paulo State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OCTGab
Record Dates: First submitted 2016-11-18; First posted 2016-11-30 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Epilepsy; Chronic Pain
Keywords: Gabapentin; OCT2; OCTN1; Pharmacogenetics; Pharmacokinetics; Polymorphisms
MeSH Terms: conditions — Epilepsy; Chronic Pain | interventions — Gabapentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Homozygous for the wild type allele (Active Comparator): Patients with 18 years old or older with epilepsy, neuropathic pain or any chronic pain undergoing chronic treatment with gabapentin are being recruited.
  Sparse blood sampling are being collected up to 4 h after administration of the drug for pharmacokinetic study. Urine sampling are being collected during the dosing interval, only in patients hospitalized at the Hospital Estadual de Américo Brasiliense (HEAB). Blood sample are being collected for DNA extraction. DNA are being extracted from the whole blood of all patients for genotyping of the SLC22A2 c.808G>T and SLC22A4 c.1507C>T polymorphisms.
  Interventions: Procedure: Sparse blood sampling; Procedure: Urine sampling; Procedure: DNA extraction; Drug: Gabapentin
- Homo- or heterozygous for rare alleles (Active Comparator): Patients with 18 years old or older with epilepsy, neuropathic pain or any chronic pain undergoing chronic treatment with gabapentin are being recruited.
  Sparse blood sampling are being collected up to 4 h after administration of the drug for pharmacokinetic study. Urine sampling are being collected during the dosing interval, only in patients hospitalized at the Hospital Estadual de Américo Brasiliense (HEAB). Blood sample are being collected for DNA extraction. DNA are being extracted from the whole blood of all patients for genotyping of the SLC22A2 c.808G>T and SLC22A4 c.1507C>T polymorphisms.
  Interventions: Procedure: Sparse blood sampling; Procedure: Urine sampling; Procedure: DNA extraction; Drug: Gabapentin

INTERVENTIONS:
Procedure: Sparse blood sampling — Blood samples are being collected at times 0, 90 and 240 minutes after gabapentin administration.
Procedure: Urine sampling — Urine samples are being collected during the dosing interval, only in patients hospitalized at Hospital Estadual de Américo Brasiliense (HEAB).
Procedure: DNA extraction — Blood sample are being collected for DNA extraction. DNA are being extracted from the whole blood of all patients for genotyping of the SLC22A2 c.808G>T and SLC22A4 c.1507C>T polymorphisms
Drug: Gabapentin — All patients undergoing chronic treatment with gabapentin are being recruited.
  Other Names: GAB

SUMMARY:
This study aims to evaluate the influence of genetic polymorphisms of OCTN1 and OCT2 and other possible covariates on the kinetic disposition of GAB in patients undergoing GAB chronic treatment. Thus, patients treated with GAB, for at least one week, are being investigated.

DETAILED DESCRIPTION:
Gabapentin (GAB), an anticonvulsant used for the treatment of epilepsy and chronic pain, has nonlinear kinetics, it is not metabolized and it is mainly eliminated by renal excretion. Studies suggest that the renal excretion of GAB is dependent on active secretion by organic cation transporter 2 (OCT2) and organic cation/ergothioneine transporter 1 (OCTN1). These transporters are expressed at the membrane of the renal proximal tubules and they are involved in the elimination of endogenous compounds and many drugs. The genetic polymorphism of drug transporters has been studied to explain the kinetic disposition variability of their substrates. The objective of this study is to investigate the influence of genetic polymorphisms of OCTN1 and OCT2 and other possible covariates (e.g., sex, age, creatinine clearance, body mass index) on the kinetic disposition of GAB in patients undergoing GAB chronic treatment. Patients treated with GAB, for at least one week, are being investigated. Blood and urine samples are being collected to GAB pharmacokinetic analysis, serum creatinine analysis and for genotyping. The plasma concentration of GAB will be assessed using liquid chromatography with UV detection (LC-UV).

ELIGIBILITY:
Inclusion Criteria:

* Patients with 18 years old or older, both gender.
* Patients undergoing chronic use of gabapentin (at least one week).

Exclusion Criteria:

* Pregnant and lactating patients.
* Patients who were in use of OCT2 and OCTN1 inhibitors.
* Patients who disagree to continue the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2016-09; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Gabapentin plasma concentration. | Up to 240 minutes after gabapentin administration.
  Blood samples will be collected at 0, 90 and 240 minutes after gabapentin administration. The gabapentin plasma concentration will be assessed using liquid chromatography with UV detection (LC-UV).
OCT2 and OCTN1 genotyping | Up to 5 minutes before gabapentin administration
  The single nucleotide polymorphisms of SLC22A2 gene (c.808G>T) and SLC22A4 (c.1507C>T) are being evaluated in all included patients.

CONTACTS AND LOCATIONS:
Overall Officials: Fabíola D. Eckeli, Prof., Principal Investigator — University of Sao Paulo; Edgar Ianhez Júnior, Principal Investigator — Hospital Estadual de Américo Brasiliense; Natália V. de Moraes, Prof., Study Chair — Universidade Estadual Paulista Júlio de Mesquita Filho
Locations (1):
- Universidade Estadual Paulista Júlio de Mesquita Filho, Araraquara, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No